CLINICAL TRIAL: NCT00184236
Title: Aerobic Interval Training Reduces Cardiovascular Risk Factors More Than a Multitreatment Approach in Overweight Adolescents
Brief Title: Cardiovascular Risk Factors in Overweight Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ts-aet01
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Overweight; Obesity
Keywords: Exercise Training; Cardiovascular diseases; Risk factors
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic interval training (Active Comparator): Aerobic interval training (AIT)
  Interventions: Behavioral: Aerobic interval training
- Multitreatment approach (Active Comparator): multitreatment approach (MTG)
  Interventions: Behavioral: Multitreatment approach

INTERVENTIONS:
Behavioral: Multitreatment approach — 12 months regimen consisting of group meetings every 2 weeks involving a physician, psychologist, physiotherapist and clinical nutritional physiologist. 21 h treatment during the first 3 months: 3 activity sessions (3 h) and 3 group conversations (4 h). Attendance inclusion criterium was set to minimum of 80%
  Other Names: multidisciplinary approach
  Arms: Multitreatment approach
Behavioral: Aerobic interval training — Walking/running 'uphill' on a treadmill twice a week for 3 months. 10 min warming-up at 70% of Hfmax before performing 4x4 intervals at 90-95% of Hfmax. 3 min active recovery at 70% of Hfmax between each interval. 5 min cool-down period, giving a total of 40 min.
  Arms: Aerobic interval training

SUMMARY:
The aim of the present study was to determine the effects of either a multidisciplinary approach or intensity-controlled interval training on cardiovascular risk factors in overweight adolescents.

DETAILED DESCRIPTION:
Several approaches have been used to improve cardiovascular health status and quality of life in obese children and adolescents, without coming to a consensus decision. Recently, a few studies have determined the effects of exercise training and diet on endothelial function in overweight and obese children and adolescents. The main findings are that only a moderate amount of exercise training and diet changes improves or restores endothelial function. It is difficult, however, to asses the separate effects of the training and diet, particularly because none of the studies have used a homogenous exercise training regimen. Unanimously, better, but affordable prevention and treatment strategies to improve wide-scale health outcome are called upon to slow down the current epidemic of overweight. It is now well established that physical activity reduces, but does not currently prevent the epidemic of obesity from either reaching global proportions or taxing public health and economy. Despite the recent advances in understanding the responsible biology of improved cardiovascular health with exercise training, several lines of research questions are still unresolved. For instance, the optimal program, e.g. when to initiate, whom to prescribe exercise to, which exercise-intensity is required, and the actual design of the treatment program, remain by far yet to determine.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese adolescents in the Trondheim area, referred to medical treatment at St. Olav's Hospital

Exclusion Criteria:

* Any coexisting medical illnesses

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
VO2max change | 3 months and 12 months
  maximal oxygen uptake change

SECONDARY OUTCOMES:
Cardiovascular risk factors | 2 years
endothelial function change | 3 months and 12 months
  measured as FMD (flow-mediated dilution) using high-resolution vascular ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, PhD prof, Study Chair — Norwegian University of Science and Technology
Locations (1):
- The Norwegian University of Science and Technology, Trondheim, Sør-Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tjonna AE, Stolen TO, Bye A, Volden M, Slordahl SA, Odegard R, Skogvoll E, Wisloff U. Aerobic interval training reduces cardiovascular risk factors more than a multitreatment approach in overweight adolescents. Clin Sci (Lond). 2009 Feb;116(4):317-26. doi: 10.1042/CS20080249. PMID 18673303
- [Result] Ingul CB, Tjonna AE, Stolen TO, Stoylen A, Wisloff U. Impaired cardiac function among obese adolescents: effect of aerobic interval training. Arch Pediatr Adolesc Med. 2010 Sep;164(9):852-9. doi: 10.1001/archpediatrics.2010.158. PMID 20819968